CLINICAL TRIAL: NCT00006265
Title: A Dose Escalation And Phase II Study Of Gemtuzumab Ozogamicin (CMA-676; Mylotarg) With High-Dose Cytarabine For Patients With Refractory Or Relapsed Acute Myeloid Leukemia (AML)
Brief Title: Gemtuzumab Ozogamicin and High-Dose Cytarabine in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-19902; U10CA031946 (NIH); CALGB-19902; CDR0000068208 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-09-11; First posted 2003-09-03 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Cytarabine; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort I (Experimental): Immunotherapy with gemtuzumab
  Interventions: Biological: gemtuzumab ozogamicin
- Cohort II (Experimental): Gemtuzumab + ara-C
  Interventions: Drug: ara-C; Biological: gemtuzumab ozogamicin
- Cohort IA (Experimental): Gemtuzumab + ara C
  Interventions: Drug: ara-C; Biological: gemtuzumab ozogamicin
- Cohort IV (Experimental): Gemtuzumab + ara-C
  Interventions: Drug: ara-C; Biological: gemtuzumab ozogamicin

INTERVENTIONS:
Drug: ara-C — 3 g/sq m IV infusion over 3 hours Days 1-5
  Other Names: Cytarabine
  Arms: Cohort IA; Cohort II; Cohort IV
Biological: gemtuzumab ozogamicin — 9 mg/sq m IV infusion over 2 hrs D 1 (Cohort I); D 7 (Cohorts II, IA, & IV); & D 14 (Cohort IV) 4.5 mg/sq m IV infusion over 2 hrs D 8 (Cohort I) & D 14 (Cohort II)
  Other Names: Mylotarg

SUMMARY:
RATIONALE: Monoclonal antibodies, such as gemtuzumab ozogamicin, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as cytarabine, use different ways to stop cancer cells from dividing so they stop growing or die. Combining gemtuzumab ozogamicin with cytarabine may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemtuzumab ozogamicin with high-dose cytarabine in treating patients who have relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with relapsed or refractory acute myeloid leukemia treated with gemtuzumab ozogamicin (CMA-676) and high-dose cytarabine.
* Determine the safety and toxicity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of gemtuzumab ozogamicin (CMA-676) (phase I closed to accrual effective 08/25/2003). Patients are stratified according to disease status (refractory vs relapsed).

* Phase I (closed to accrual effective 08/25/2003): Patients are enrolled in one of four cohorts.

  * Cohort I (closed to accrual as of 10/1/02): Patients receive CMA-676 at the first dose level IV over 2 hours on days 1 and 8.
  * Cohort IA (open to accrual as of 10/15/02): Patients receive high-dose cytarabine (HD-ARA-C) IV over 3 hours on days 1-5 and CMA-676 IV over 2 hours on day 7.
  * Cohort II: Patients receive HD-ARA-C as in cohort IA and CMA-676 at the first dose level IV over 2 hours on days 7 and 14.
  * Cohort IV: Patients receive CMA-676 at the second dose level and HD-ARA-C as in cohort II.

Dose escalation stops if at least 3 of 9 patients experience dose-limiting toxicity.

* Phase II: Patients receive HD-ARA-C IV over 3 hours on days 1-5 and CMA-676 IV over 2 hours on day 7 (one course).

Patients are followed at 1 month, monthly for 6 months, every 3 months for 2 years, and then annually for 10 years.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for phase I of the study and a total of 37 patients will be accrued for phase II of the study within 2 years. (Phase I closed to accrual effective 08/25/2003).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Primary refractory acute myeloid leukemia (AML)

    * More than 10% blasts in the bone marrow or blood after recovery from 2 courses of standard cytarabine- and anthracycline-based induction chemotherapy
    * No prior remission
  * Relapsed AML

    * More than 10% blasts in the bone marrow or blood after documented remission
    * Prior remission lasted more than 30 days
    * No prior treatment for current relapse
* CD33 expression on at least 20% of leukemia blast cells at initial diagnosis for primary refractory patients or at the time of relapse for all other patients
* No active CNS involvement

PATIENT CHARACTERISTICS:

Age:

* 17 and over

Performance status:

* 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* WBC less than 30,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* No veno-occlusive disease of the liver
* No chronic liver disease unless due to AML

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active serious infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 6 months since prior stem cell transplantation

Chemotherapy:

* See Disease Characteristics
* Prior etoposide and/or thioguanine during remission induction allowed
* Prior hydroxyurea for control of AML allowed
* At least 24 hours since prior hydroxyurea
* At least 3 months since prior high-dose cytarabine (greater than 2 g/m^2/dose)-containing regimen
* No other concurrent chemotherapy

Endocrine therapy:

* Concurrent steroids for adrenal failure, hypersensitivity reactions, or septic shock allowed
* Concurrent ophthalmic corticosteroids allowed
* Concurrent hormones for nondisease-related conditions (e.g., insulin for diabetes or estrogens or progestins for gynecologic conditions) allowed

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* More than 2 months since prior cytotoxic therapy

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2001-03; Primary Completion 2004-12 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Complete remission rate | 8 or 14 days after tx initiation & 30 d post tx

SECONDARY OUTCOMES:
Toxicity | D 14, then 30, 60 , & 90 d post Tx, q 3 mon for 1 yr, then at relapse or death

CONTACTS AND LOCATIONS:
Overall Officials: Richard Stone, MD, Study Chair — Dana-Farber Cancer Institute
Locations (78):
- United States (77):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth Medical School, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Oklahoma University Medical Center at University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico

REFERENCES:
- [Result] Stone RM, Moser B, Sanford B, Schulman P, Kolitz JE, Allen S, Stock W, Galinsky I, Vij R, Marcucci G, Hurd D, Larson RA; Cancer and Leukemia Group B. High dose cytarabine plus gemtuzumab ozogamicin for patients with relapsed or refractory acute myeloid leukemia: Cancer and Leukemia Group B study 19902. Leuk Res. 2011 Mar;35(3):329-33. doi: 10.1016/j.leukres.2010.07.017. Epub 2010 Aug 4. PMID 20688393
- [Result] Stone RM, Moser B, Schulman P, et al.: A dose escalation and phase II study of gemtuzumab ozogamicin (GO) with high-dose cytarabine (HiDAC) for patients (pts) with refractory or relapsed acute myeloid leukemia (AML): CALGB 19902. [Abstract] Blood 104 (11): A-873, 2004.